CLINICAL TRIAL: NCT06144905
Title: Gut Microbiota Alterations in Anorexia Nervosa - Paving the Way for Personalized Prebiotic Treatment Strategies
Brief Title: Norwegian Microbiota Study in Anorexia Nervosa
Acronym: NORMA
Status: Recruiting | Type: Observational
Sponsor: Norwegian University of Life Sciences (Other)
Collaborators: Oslo University Hospital (Other); Helse Nord-Trøndelag HF (Other); Haukeland University Hospital (Other); Nordlandssykehuset HF (Other); Modum Bad (Other); Karolinska Institutet (Other); The Eating disorder Association, Norway (SPISFO) (Unknown); Counseling on eating disorders, Norway (ROS) (Unknown)
Responsible Party: Principal Investigator, Siv K Bohn, Professor, Norwegian University of Life Sciences
Other Study IDs: 336239_KBM_SKB2023
Record Dates: First submitted 2023-09-22; First posted 2023-11-22 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Anorexia Nervosa; Mental Health Issue; Microbiota; Diet; Gastrointestinal Problems
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Fecal samples for microbiota investigation and serum samples will be collected at several time points for the patients with anorexia nervosa: 1) before admission to the hospital, 2, after about 6 weeks and 3) after about 12 weeks. For the control group the biospecimen will be collected at one time-point only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Anorexia nervosa (AN) group: Female in-patients with anorexia nervosa, age 16-50 years with BMI below 18.5 kg/m2.
  Interventions: Other: standard care treatment program
- Heathy control (HC) group: Female healthy controls, age 16-50 with normal to mild overweight (18.5 ≤ BMI< 27 kg/m2). .

INTERVENTIONS:
Other: standard care treatment program — The standard care treatment consists of a program of psychotherapy and nutritional rehabilitation to achieve normalization of food-intake and weight gain.
  Groups: Anorexia nervosa (AN) group

SUMMARY:
Anorexia nervosa (AN) is a serious mental disorder occurring mainly in women. AN is characterized by severely restricted food-intake and subsequent low weight. The disease burden for the individual is high with medical complications and psychiatric comorbidities. Despite decades of research, there are large gaps in the understanding of the biological aspects of AN and lack of effective interventions. Current clinical treatment is associated with gastrointestinal problems, high rates of relapse and poor outcome causing long-term sickness absence and disability. During the COVID19 pandemic the prevalence and severity of AN has spiked. Therefore, there is great need of novel strategies for AN treatment, that can be easily implemented in the clinic without adding complexity to the standard care of treatment. During the resent years it has been proposed that mental disorders might be treated via manipulating the composition and function of the microbes that live in the gut (the microbiota) by adding or restricting fermentable nutrients (prebiotics) in the diet. However, in order to use prebiotics to treat the microbiota in AN patients, more knowledge is needed on how the AN microbiota is affected by the current standard care treatment. Whether prebiotics can be useful for normalizing AN microbiota remains to be established. The overall aim of the "Norwegian study of Microbiota in Anorexia Nervosa" (NORMA) is to join forces of researchers, clinical health care services and voluntary sector in a transdiciplinary approach to improve the understanding of the role of the gut microbiota in AN patients. The current project will include a clinical trial in AN patients and experimental studies to screen novel prebiotics for their ability to modify and normalize AN derived microbiota. The long-term goal of the project is to pave the way for a targeted and clinically feasible individualized treatment for better tolerable weight-restoration and improved health in AN patients.

ELIGIBILITY:
Inclusion Criteria AN group

1. Sex: Female
2. Age: 16-50 years
3. BMI: <18.5 kg/m2
4. fulfilling ICD-10 criteria for AN
5. currently referred to specialized inpatient nutritional treatment for AN
6. able to understand the Norwegian questionnaires.

Exclusion Criteria AND group:

1. history of inflammatory bowel disease, celiac disease, or GI tract surgery;
2. treatment with oral antibiotics the past two months
3. high intake of probiotic supplements over the past two months.

Inclusion criteria control group

1. Sex: Female
2. Age: 16-50 years
3. BMI: >= 18.5 & < 27
4. able to understand the Norwegian questionnaires.

Exclusion Criteria AND group:

1. history of inflammatory bowel disease, celiac disease, or GI tract surgery;
2. treatment with oral antibiotics the past two months
3. high intake of probiotic supplements over the past two months.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: The female patients with anorexia nervosa (AN) are undergoing specialized nutritional rehabilitation treatment and will be recruited from five Norwegian specialized inpatient treatment units for eating disorders. The standard care treatment consists of a program of psychotherapy and nutritional rehabilitation to achieve normalization of food-intake and weight gain. Although the clinical strategy of AN treatment is standardized, both the psychotherapy and dietary advices are individualized. The dietary advice during standard care treatment is based on clinical experience, as specific guidelines are lacking. Diets are adapted to each individual in aspects of tolerability and preferences, but typically comprise a high-energy diets aiming for a weekly weight gain of 0.5-1.5 kilograms. Often enteral nutrition (i.e., tube feeding) is required. The control group will be aged-matched female subjects with normal weight - mildly overweight.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-09-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2043-09 (Estimated)

PRIMARY OUTCOMES:
Differences in the fecal microbiota composition | Cross-sectional study with only one time point. For AN-group; the baseline sample is delivered during the last week before start of clinical treatment. ]
  Comparison of fecal microbial composition between the patients with anorexia nervosa and healthy controls. We will compare different indices of α-diversity - investigating both richness and evenness (e.g. observed number of OTUs, Chao1, Shannon-Wiener, Simpson, and PD whole tree) and different indices of β-diversity (e.g. binary Jaccard, Bray-Curtis, and weighted Unifrac). Also differences in bacterial abundances at various taxonomic levels (phylum, class, order, family, and genus) will be investigated.
Change in the fecal microbiota composition in patients with anorexia nervosa during the standard care treatment at the clinics for eating disorder. | One group time-series design. Samples will be taken at baseline (~one week before admission to the clinic) and at ~6 weeks and ~12 weeks.
  Mixed model analyses will be performed to assess whether the standard care treatment at the clinics for eating disorder induce changes in the fecal microbiota composition. Both diversity measures ( α-diversity and β-diversity) and bacterial abundances at various taxonomic levels (phylum, class, order, family, and genus) will be investigated.
Change in mental scores during standard care treatment at the clinics for eating disorder | One group time-series design. Data will be collected at baseline, at admission to the clinic and at ~6 weeks and ~12 weeks.
  Mixed model analyses will be performed to assess whether the standard care treatment at the clinics for eating disorder induce changes in mental scores. Effects of time will be investigated in the AN group only. Mental scores will be assessed using digital questionnaires.
Change in gastrointestinal problems during standard care treatment at the clinics for eating disorder | One group time-series design. Data will be collected at baseline, at admission to the clinic and at ~6 weeks and ~12 weeks.
  Mixed model analyses will be performed to assess whether the standard care treatment at the clinics for eating disorder induce changes in gastrointestinal problems. Effects of time will be investigated in the AN group only. Scores for gastrointestinal problems will be assessed using digital questionnaires.

SECONDARY OUTCOMES:
Associations between microbiota measures (diversity and abundance of specific species), serum biomarkers, dietary charachteristics, gastrointestinal issues and mental issues. | Cross-sectional study with only one time point. For AN-group; the baseline sample is delivered during the last week before start of clinical treatment. ]
  Associations between multiple variables will be investigated in both AN group (at baseline, 6 weeks and 12 weeks) and HC group at baseline using unsupervised learning algorithm techniques such as Principal Component Analysis and hireachical clustering techniques. Microbiota is charachterized as described under outcome 1, serum biomarkers include standard clinical biomarkers and biomarkers of inflammation and microbiota relevant biomarkers. Data on dietary charachteristics, gastrointestinal issues and mental issues are obtained by digital questionnaires.
Associations between baseline microbiota composition and changes in gastrointestinal complaints during the standard care treatment at the clinics for eating disorder. | One group time-series design. Samples, data will be obtained at baseline (~one week before admission to the clinic) and at ~6 weeks and ~12 weeks.
  Associations between microbiota measures at baseline and changes in gastrointestinal complaint sduring the standard care treatment at the clinics for eating disorder will be investigated by unsupervised learning algorithm techniques such as Principal Component Analysis and by applying hireachical clustering techniques on correlation measures. Microbiota will be charachterized as described under outcome 1, serum biomarkers include standard clinical biomarkers and biomarkers of inflammation and microbiota relevant biomarkers. Data on dietary charachteristics, gastrointestinal issues and mental issues are obtained by digital questionnaires.
Associations between baseline microbiota composition and changes in mental scores during the standard care treatment at the clinics for eating disorder. | One group time-series design. Samples, data will be obtained at baseline (~one week before admission to the clinic) and at ~6 weeks and ~12 weeks.
  Associations between microbiota measures at baseline and changes in mental scores during the standard care treatment at the clinics for eating disorder will be investigated by unsupervised learning algorithm techniques such as Principal Component Analysis and by applying hireachical clustering techniques on correlation measures. Microbiota will be charachterized as described under outcome 1, serum biomarkers include standard clinical biomarkers and biomarkers of inflammation and microbiota relevant biomarkers. Data on dietary charachteristics, gastrointestinal issues and mental issues are obtained by digital questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Siv K Bøhn, PhD, Principal Investigator — Norwegian University of Life Sciences
Locations (1):
- Norwegian University of Life Sciences, Ås, Ås, Norway

IPD SHARING:
Plan to Share IPD: Undecided